CLINICAL TRIAL: NCT04669067
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of TL-895 Combined With KRT-232 in Patients With Relapsed/Refractory (R/R) FLT3+ Acute Myeloid Leukemia (AML)
Brief Title: TL-895 and KRT-232 Study in Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Telios Pharma, Inc. (Industry)
Collaborators: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL-895-203
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; TP53; FLT3+; Navtemadlin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b - Dose Level 1 (Experimental): KRT-232 240mg QD, orally administered on days 1 through 7 of each 28-day cycle in combination with TL-895 150mg BID continuously for each 28-day cycle.
  Interventions: Drug: TL-895; Drug: KRT-232
- Phase 1b - Dose Level 2 (Experimental): KRT-232 300mg QD, orally administered on days 1 through 7 of each 28-day cycle in combination with TL-895 150mg BID continuously for each 28-day cycle.
  Interventions: Drug: TL-895; Drug: KRT-232
- Phase 1b - Dose Level 3 (Experimental): Cycle 1 only: KRT-232 360 mg QD orally administered on Days 1 through 7 of the first 28-day cycle in combination with TL-895 150 mg BID continuously for the first 28-day cycle
  Cycle 2 and beyond: KRT-232 300 mg QD orally administered on Days 1 through 7 of each 28-day cycle in combination with TL-895 150 mg BID continuously for each 28-day cycle.
  Interventions: Drug: TL-895; Drug: KRT-232
- Phase 1b - Dose Level 4 (Experimental): Cycle 1 only: KRT-232 360 mg QD orally administered on Days 1 through 7 of the first 28-day cycle in combination with TL-895 300 mg BID continuously for the first 28-day cycle.
  Cycle 2 and beyond: KRT-232 300 mg QD orally administered on Days 1 through 7 of each 28-day cycle in combination with TL-895 300 mg BID continuously for each 28-day cycle.
  Interventions: Drug: TL-895; Drug: KRT-232
- Phase 1b - Dose Level 5 (Experimental): Cycle 1 only: KRT-232 360 mg QD orally administered on Days 1 through 7 of the first 28-day cycle in combination with TL-895 450 mg BID continuously for the first 28-day cycle.
  Cycle 2 and beyond: KRT-232 300 mg QD orally administered on Days 1 through 7 of each 28-day cycle in combination with TL-895 450 mg BID continuously for each 28-day cycle.
  Interventions: Drug: TL-895; Drug: KRT-232
- Phase 2 - Dose Expansion (Experimental): Dose expansion of the recommended phase 2 dose of TL-895 in combination with KRT-232 as determined in Phase 1b.
  Interventions: Drug: TL-895; Drug: KRT-232

INTERVENTIONS:
Drug: TL-895 — TL-895 is an experimental tyrosine kinase inhibitor anticancer drug taken by mouth.
Drug: KRT-232 — KRT-232 is an experimental MDM2 inhibitor anticancer drug taken by mouth.

SUMMARY:
This study evaluates TL-895, a potent, orally available and highly selective irreversible tyrosine kinase inhibitor combined with navtemadlin (KRT-232), a novel oral small molecule inhibitor of MDM2 for the treatment of adults with FLT3 mutated Acute Myeloid Leukemia. Participants must be relapsed/refractory (e.g., having failed prior therapy) to be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* TP53 wildtype AML
* Relapsed/Refractory to at least one prior therapy, one of which must have included a FLT-3 inhibitor
* FLT3 mutation (FLT3-TKD or FLT3-ITD)
* ECOG 0-2
* Adequate hematologic, hepatic, and renal functions

Exclusion Criteria:

* AML subtype 3
* Prior treatment with MDM2 antagonist therapies
* Eligible for HSCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Primary Objective, Phase 1b: To determine the MTD/MAD and recommended Phase 2 dose (RP2D) of TL-895 in combination with KRT-232 | 13 months
  Dose limiting toxicities will be used to established the MTD/MAD of TL-895 combined with KRT-232. The Safety Review Committee (SRC) will determine the RP2D based on safety data of the combination of TL-895 and KRT-232.
Primary Objective, Phase 2: To determine the rates of complete remission (CR) and complete remission with partial hematologic recovery (CRh) | 41 months
  The proportion of subjects who achieved CR or CRh as their best response based on the Modified 2017 European LeukemiaNet (ELN) Response Criteria (Appendix 4).

SECONDARY OUTCOMES:
Key Secondary Objective: To determine the overall response rate (ORR) | 41 months
  The proportion of subjects who achieve PR or better.
Key Secondary Objective: To determine the duration of CR/CRh response (DOR) | 41 months
  Median DOR (Kaplan-Meier estimate) defined as the time from first observation of CR/CRh to relapse or death from any cause, whichever occurs first. Subjects with MLFS by bone marrow biopsy performed earlier in the course of therapy who convert to CR or CRh do not require a separate bone marrow aspirate at the time of CR or CRh to document this.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (11):
  - Keck School of Medicine, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Georgia Cancer Center, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Division of Hematology Oncology and Cell Therapy, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weill Cornell Medical College, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Research Organization, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Harold C. Simmons Cancer Center, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - University of Sunshine Coast-Sippy Downs, Sippy Downs
  - Westmead Hospital, Sydney
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Medical University Vienna, Department of Internal Medicine I, Clinical Department of Hematology and Hemostaseology, Vienna
- France (6):
  - Claude Huriez Hospital, Lille
  - South Lyon Hospital Center, Lyon
  - Paoli-Calmettes Institute, Marseille
  - University Hospital of Nantes, Nantes
  - Hospital Center Universitaire De Nice, Nice
  - Saint-Louis Hospital, Paris
- Germany (5):
  - University Hospital Halle (Saale), Department of Internal Medicine IV - Hematology and Oncology, Halle, Saxony-Anhalt
  - University Duisburg-Essen, University Hospital Essen, Department of Internal Medicine, Essen
  - University Hospital Hamburg-Eppendorf, Department of Internal Medicine II, Hamburg
  - Hannover Medical School, Center for Internal Medicine, Clinic of Hematology, Hemostaseology, Oncology and Stem Cell Transplantation, Hanover
  - University Hospital Jena, Clinic of Internal Medicine II, Department of Hematology and Medical Oncology, Jena
- Italy (3):
  - University Hospital - Ospedali Riuniti Umberto I - GM Lancisi - G Salesi of Ancona, Haematology Clinic, Ancona
  - Polyclinic S. Orsola-Malpighi, Operative Unit of Hematology, Bologna
  - Romagnolo Scientific Institute of Meldola (IRST) S.r.l., Department of Oncology and Clinical and Experimental Haematology, Meldola
- South Korea (2):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Department of Hemato-Oncology, Seoul
- Spain (4):
  - University Hospital Germans Trias i Pujol, Department of Clinical Hematology, Badalona
  - University Hospital Vall d'Hebron, Barcelona
  - University Clinical Hospital of Valencia, Department of Hematology and Medical Oncology, Valencia
  - Hospital Universitario y Politécnico de La Fe, Valencia